CLINICAL TRIAL: NCT00463866
Title: Local Phase 4 Pan-European SMART Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5890L00022; EUROSMART; EudraCTNo. 2006-006512-30
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Results first posted 2010-03-22 (Estimated); Last update posted 2010-03-22 (Estimated); Status verified 2010-03

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination

INTERVENTIONS:
Drug: Budesonide/formoterol

SUMMARY:
The purpose of this study is to evaluate the effect of two different maintenance doses of Symbicort Maintenance And Reliever Therapy (SMART) in adult asthmatic patients. A 6 month treatment period

ELIGIBILITY:
Inclusion Criteria:

* Patients at out-patient clinics
* >18 years with a minimum of 6 months documented history of persistent asthma who have used inhaled glucocorticosteroids for at least one month and have a history of use in rapid-acting B2 agonists for symptom relief

Exclusion Criteria:

* Asthma exacerbation within the last 14 days prior to study start
* subject aged >40 years with a smoking history of >10pack-years
* subjects with chronic obstructive lung disease or other significant respiratory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8424 (Actual)
Dates: Start 2007-03; Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Aubier, Prof, Principal Investigator — FRANCE; Juliette Ostinelli, MD, Study Chair — AstraZeneca, MC France
Locations (817):
- Belgium (125):
  - Research Site, Aalst
  - Research Site, Aarschot
  - Research Site, Aatrijken
  - Research Site, Asse
  - Research Site, Balen
  - Research Site, Bastogne
  - Research Site, Bellaire
  - Research Site, Betrix
  - Research Site, Binche
  - Research Site, Blankenberge
  - Research Site, Boortmeerbeek
  - Research Site, Bornem
  - Research Site, Boussu
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Buizingen
  - Research Site, Burdinne
  - Research Site, Champion
  - Research Site, Charleroi
  - Research Site, Châtelet
  - Research Site, Chênée
  - Research Site, Dendermonde
  - Research Site, Diksmuide
  - Research Site, Drongen
  - Research Site, Duffel
  - Research Site, Edegem
  - Research Site, Eeklo
  - Research Site, Ekeren
  - Research Site, Erembodegem
  - Research Site, Evergem
  - Research Site, Fleurus
  - Research Site, Gembloux
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Gilly
  - Research Site, Graty
  - Research Site, Grivegnée
  - Research Site, Halle
  - Research Site, Ham
  - Research Site, Ham-sur-Heure
  - Research Site, Hasselt
  - Research Site, Havinnes
  - Research Site, Heist-op-den-Berg
  - Research Site, Herentals
  - Research Site, Herstal
  - Research Site, Hoboken
  - Research Site, Hoeselt
  - Research Site, Hooglede
  - Research Site, Hornu
  - Research Site, Houthalen-Helchteren
  - Research Site, Huldenberg
  - Research Site, Izegem
  - Research Site, Jambes
  - Research Site, Jodoigne
  - Research Site, Kinrooi
  - Research Site, Kontich
  - Research Site, Kraainem
  - Research Site, La Louvière
  - Research Site, Langdorp
  - Research Site, Lauwe
  - Research Site, Leopoldsburg
  - Research Site, Leuven
  - Research Site, Lier
  - Research Site, Liège
  - Research Site, Lommel
  - Research Site, Lovendegem
  - Research Site, Malmedy
  - Research Site, Marchovelette
  - Research Site, Meelbeke
  - Research Site, Moerkerke
  - Research Site, Mol
  - Research Site, Monceau-sur-Sambre
  - Research Site, Mons
  - Research Site, Montegnée
  - Research Site, Moorsel
  - Research Site, Mouscron
  - Research Site, Namur
  - Research Site, Natoye
  - Research Site, Nijlen
  - Research Site, Nivelles
  - Research Site, Oedelem
  - Research Site, Oostkamp
  - Research Site, Oppuurs
  - Research Site, Ostend
  - Research Site, Oudenaarde
  - Research Site, Paal
  - Research Site, Peutie
  - Research Site, Poederlee
  - Research Site, Pulle
  - Research Site, Rijkevorsel
  - Research Site, Rixensart
  - Research Site, Rotselaar
  - Research Site, Roux
  - Research Site, Saint Katharina Lombeek
  - Research Site, Sankt Vith
  - Research Site, Sijsele
  - Research Site, Sint-Genesius-Rode
  - Research Site, Sint-Niklaas
  - Research Site, Steenokkerzeel
  - Research Site, Stekene
  - Research Site, Tavier
  - Research Site, Thieusies
  - Research Site, Tielt
  - Research Site, Tienen
  - Research Site, Tirlt
  - Research Site, Tongeren
  - Research Site, Tournai
  - Research Site, Tremelo
  - Research Site, Turhout
  - Research Site, Vedrin
  - Research Site, Villers-Poterie
  - Research Site, Vilvoorde
  - Research Site, Vosselaar
  - Research Site, Wambeek
  - Research Site, Waregem
  - Research Site, Waterloo
  - Research Site, Wetteren
  - Research Site, Wijnegem
  - Research Site, Willebroek
  - Research Site, Wilsele
  - Research Site, Zele
  - Research Site, Zemst
  - Research Site, Zoersel
  - Research Site, Zottegem
  - Research Site, Zwijnaarde
- Finland (43):
  - Research Site, Espho
  - Research Site, Espoo
  - Research Site, Harjavalta
  - Research Site, Hämeenlinna
  - Research Site, Helsinki
  - Research Site, Hyvinkää
  - Research Site, Jakobstad
  - Research Site, Joensuu
  - Research Site, Jokioinen
  - Research Site, Kannus
  - Research Site, Kemi
  - Research Site, Kereva
  - Research Site, Kokkola
  - Research Site, Korpilahti
  - Research Site, Kotka
  - Research Site, Kouvola
  - Research Site, Kuopio
  - Research Site, Kuusankoski
  - Research Site, Lahti
  - Research Site, Lappeenranta
  - Research Site, Lapua
  - Research Site, Lathi
  - Research Site, Lempäälä
  - Research Site, Lohja
  - Research Site, Mikkeli
  - Research Site, Muurame
  - Research Site, Nurmij�rvi
  - Research Site, Oulu
  - Research Site, Pello
  - Research Site, Pieksämäki
  - Research Site, Pori
  - Research Site, Porvoo
  - Research Site, Pudasj�rvi
  - Research Site, Pyhäjoki
  - Research Site, Riihimäki
  - Research Site, Seinäjoki
  - Research Site, Suonenjoki
  - Research Site, Tamepare
  - Research Site, Tampera
  - Research Site, Turku
  - Research Site, Ulvila
  - Research Site, Vaajakoksi
  - Research Site, Vantaa
- France (184):
  - Research Site, Agen
  - Research Site, Aix-en-Provence
  - Research Site, Ajaccio
  - Research Site, Alès
  - Research Site, Amboise
  - Research Site, Amelie Les Bains Palalda
  - Research Site, Amiens
  - Research Site, Angers
  - Research Site, Angoulême
  - Research Site, Annecy
  - Research Site, Annonay
  - Research Site, Antibes
  - Research Site, Arpajon
  - Research Site, Asnières-sur-Seine
  - Research Site, Aubagne
  - Research Site, Aulnay-sous-Bois
  - Research Site, Avignon
  - Research Site, Bastia
  - Research Site, Bayonne
  - Research Site, Belfort
  - Research Site, Bernay
  - Research Site, Besançon
  - Research Site, Béthune
  - Research Site, Béziers
  - Research Site, Biganos
  - Research Site, Bois-Guillaume
  - Research Site, Bordeaux
  - Research Site, Bouoin Jallieu
  - Research Site, Bourges
  - Research Site, Brest
  - Research Site, Briey
  - Research Site, Brive-la-Gaillarde
  - Research Site, Cachan
  - Research Site, Caen
  - Research Site, Cagnes-sur-Mer
  - Research Site, Caluire-et-Cuire
  - Research Site, Cambrai
  - Research Site, Carpentras
  - Research Site, Castelnau-le-Lez
  - Research Site, Castres
  - Research Site, Cavaillon
  - Research Site, Challans
  - Research Site, Charleville-Mézières
  - Research Site, Chauny
  - Research Site, Chaville
  - Research Site, Châlons-en-Champagne
  - Research Site, Châteauroux
  - Research Site, Chevillu Larue Cedex
  - Research Site, Cholet
  - Research Site, Cluses
  - Research Site, Colmar
  - Research Site, Colma
  - Research Site, Colomiers
  - Research Site, Corbeil-Essonnes
  - Research Site, Créteil
  - Research Site, Denain
  - Research Site, Eaubonne
  - Research Site, Échirolles
  - Research Site, Écully
  - Research Site, Épernay
  - Research Site, Épinal
  - Research Site, Étampes
  - Research Site, Férolles-Attilly
  - Research Site, Forbach
  - Research Site, Gentilly
  - Research Site, Gleizé
  - Research Site, Grasse
  - Research Site, Grenoble
  - Research Site, Hagondange
  - Research Site, Hazebrouck
  - Research Site, Herblay-sur-Seine
  - Research Site, Hyères
  - Research Site, Joué-lès-Tours
  - Research Site, Juan-les-Pins
  - Research Site, La Garda
  - Research Site, La Roche-sur-Yon
  - Research Site, La Rochelle
  - Research Site, La Teste-de-Buch
  - Research Site, Lagny-sur-Marne
  - Research Site, Langon
  - Research Site, Laval
  - Research Site, Le Bouscat
  - Research Site, Le Perreux-sur-Marne
  - Research Site, Lens
  - Research Site, Les Sbles D Olonne
  - Research Site, Libourne
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lorient
  - Research Site, Lunel
  - Research Site, Lunéville
  - Research Site, Lyon
  - Research Site, Maisons-Laffitte
  - Research Site, Mandelieu-la-Napoule
  - Research Site, Marmande
  - Research Site, Marseille
  - Research Site, Marselle
  - Research Site, Martigues
  - Research Site, Maubeuge
  - Research Site, Meaux
  - Research Site, Melun
  - Research Site, Mende
  - Research Site, Menton
  - Research Site, Metz
  - Research Site, Montauban
  - Research Site, Montbéliard
  - Research Site, Montereau-Fault-Yonne
  - Research Site, Montferrier-sur-Lez
  - Research Site, Montigny-lès-Metz
  - Research Site, Montpellier
  - Research Site, Montreuil
  - Research Site, Nantes
  - Research Site, Narbonne
  - Research Site, Nevers
  - Research Site, Nice
  - Research Site, Niort
  - Research Site, Nîmes
  - Research Site, Obernai
  - Research Site, Ollioules
  - Research Site, Oloron-Sainte-Marie
  - Research Site, Orange
  - Research Site, Orléans
  - Research Site, Oyonnax
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Perpignan
  - Research Site, Pertuis
  - Research Site, Périgueux
  - Research Site, Pézenas
  - Research Site, Poitiers
  - Research Site, Pontault-Combault
  - Research Site, Pontoise
  - Research Site, Privas
  - Research Site, Quimper
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Rezé
  - Research Site, Roanne
  - Research Site, Rochefort
  - Research Site, Romans-sur-Isère
  - Research Site, Romorantin-Lanthenay
  - Research Site, Rosny-sous-Bois
  - Research Site, Rouen
  - Research Site, Rueil-Malmaison
  - Research Site, Saint Andre Les Verges
  - Research Site, Saint Orenes de Gameville
  - Research Site, Saint-Amand-les-Eaux
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Denis
  - Research Site, Saint-Dizier
  - Research Site, Saint-Estève
  - Research Site, Saint-Etienne
  - Research Site, Saint-Girons
  - Research Site, Saint-Herblain
  - Research Site, Saint-Jean-de-Luz
  - Research Site, Saint-Jean-de-Maurienne
  - Research Site, Saint-Laurent-du-Var
  - Research Site, Saint-Quentin
  - Research Site, Saint-Raphaël
  - Research Site, Saintes
  - Research Site, Salon-de-Provence
  - Research Site, Sarlat La Ceneda
  - Research Site, Schiltigheim
  - Research Site, Sedan
  - Research Site, Sélestat
  - Research Site, Six-Fours-les-Plages
  - Research Site, St-Malo
  - Research Site, St.-Jean
  - Research Site, Ste Feyre
  - Research Site, Strasbourg
  - Research Site, Tergnier
  - Research Site, Thionville
  - Research Site, Thonon-les-Bains
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Valence
  - Research Site, Vannes
  - Research Site, Verneuil-sur-Seine
  - Research Site, Vienne
  - Research Site, Villebon-sur-Yvette
  - Research Site, Villejuif
  - Research Site, Viooefranche Sur Saone
  - Research Site, Voiron
- Germany (130):
  - Research Site, Aachen
  - Research Site, Annaberg-Buchholz
  - Research Site, Ansbach
  - Research Site, Apolda
  - Research Site, Aschaffenburg
  - Research Site, Auerbach
  - Research Site, Augusburg
  - Research Site, Bad Bramstedt
  - Research Site, Bad Lippspringe
  - Research Site, Bad Naustadt
  - Research Site, Bad Sassendorf
  - Research Site, Bergkamen
  - Research Site, Bergrheinfeld
  - Research Site, Berlin
  - Research Site, Bernau
  - Research Site, Bernsheim
  - Research Site, Beucha
  - Research Site, Bochum
  - Research Site, Bockenem
  - Research Site, Bogen
  - Research Site, Bonn
  - Research Site, Borna
  - Research Site, Braunschweig
  - Research Site, Buchholz
  - Research Site, Burgwedel
  - Research Site, Chemnitz
  - Research Site, Cologne
  - Research Site, Coswig
  - Research Site, Cottbus
  - Research Site, Deggendorf
  - Research Site, Dillingen
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Emeden
  - Research Site, Eppelborn
  - Research Site, Erfurt
  - Research Site, Essen
  - Research Site, Esslingen am Neckar
  - Research Site, Flensburg
  - Research Site, Frankfurt
  - Research Site, Freiberg
  - Research Site, Freital
  - Research Site, Fürstenfeldbruck
  - Research Site, Fürstenwalde
  - Research Site, Fürth
  - Research Site, Geesthacht
  - Research Site, Geisen
  - Research Site, Gelnhausen
  - Research Site, Gelsenkirchen
  - Research Site, Greven
  - Research Site, Gütersloh
  - Research Site, Hagen
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Heilbronn
  - Research Site, Hsloch
  - Research Site, Ingolstadt
  - Research Site, Kaarst
  - Research Site, Karlsruhe
  - Research Site, Karlsruhe-Durlach
  - Research Site, Kassel
  - Research Site, Katzhütte
  - Research Site, Kempten
  - Research Site, Ketzin
  - Research Site, Kiel
  - Research Site, Kippenheim
  - Research Site, Kirchhain
  - Research Site, Krefeld
  - Research Site, Laage
  - Research Site, Landsberg
  - Research Site, Lebach
  - Research Site, Leipzig
  - Research Site, Lippstadt
  - Research Site, Lübeck
  - Research Site, Lüdenscheid
  - Research Site, Lütjenburg
  - Research Site, Magdenburg
  - Research Site, Mainz
  - Research Site, Marburg
  - Research Site, Marl
  - Research Site, Meisen
  - Research Site, Mittelbach
  - Research Site, Moers
  - Research Site, Mühlhausen
  - Research Site, Mülheim
  - Research Site, Mülsen
  - Research Site, München
  - Research Site, Neukirchen-Vluyn
  - Research Site, Neunkirchen
  - Research Site, Neunstadt
  - Research Site, Neuss
  - Research Site, Niesky
  - Research Site, Oranienburg
  - Research Site, Oschersleben
  - Research Site, Osnabr�ck
  - Research Site, Pirmasens
  - Research Site, Potsdam
  - Research Site, Potsda
  - Research Site, Rathenow
  - Research Site, Ratingen
  - Research Site, Recklinghausen
  - Research Site, Remscheid
  - Research Site, Rodgau
  - Research Site, Saarbrücken
  - Research Site, Saarlouis
  - Research Site, Sangerhausen
  - Research Site, Schimiedeberg
  - Research Site, Schwetzingen
  - Research Site, Silbitz
  - Research Site, Sindelfingen
  - Research Site, Solingen
  - Research Site, Stade
  - Research Site, Steinhagen
  - Research Site, Stockach
  - Research Site, Straelen
  - Research Site, Stutensee
  - Research Site, Stuttgart
  - Research Site, Tiefenbach
  - Research Site, Ueckermünde
  - Research Site, Wallerfangen
  - Research Site, Wedel
  - Research Site, Weimar
  - Research Site, Wesseling
  - Research Site, Weyhe
  - Research Site, Wilhelmshaven
  - Research Site, Wunstorf
  - Research Site, Wuppertal
- Greece (6):
  - Research Site, Alexandroupolos
  - Research Site, Athens
  - Research Site, Crete
  - Research Site, Kavala
  - Research Site, Larissa
  - Research Site, Thessaloniki
- Research Site, Reykjavik, Iceland
- Ireland (24):
  - Research Site, Bautry
  - Research Site, Beaumont Park
  - Research Site, Bishopstown
  - Research Site, Blaemy
  - Research Site, Blanchardstown
  - Research Site, Canigtwohill
  - Research Site, Carlow Town
  - Research Site, Carrigaline
  - Research Site, Clonakilty
  - Research Site, Douglas East
  - Research Site, Drogheda
  - Research Site, Dublin
  - Research Site, Gorey
  - Research Site, Headford
  - Research Site, Kilfinanen
  - Research Site, Kilmallock
  - Research Site, Kinvarra
  - Research Site, Macroom
  - Research Site, Mallow
  - Research Site, Maynooth
  - Research Site, Mullingar
  - Research Site, Naas
  - Research Site, Phibsborough
  - Research Site, Wexfoord
- Italy (76):
  - Research Site, Acquaviva Della Fonti
  - Research Site, Alba
  - Research Site, Alessandria
  - Research Site, Arezzo
  - Research Site, Ascoli Piceno
  - Research Site, Avellino
  - Research Site, Bari
  - Research Site, Benevento
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Busto Arsizio
  - Research Site, Cagliari
  - Research Site, Cantanzaro
  - Research Site, Caserta
  - Research Site, Catania
  - Research Site, Catanzaro
  - Research Site, Cattinara
  - Research Site, Cava de' Tirreni
  - Research Site, Chieti
  - Research Site, Cittadella
  - Research Site, Como
  - Research Site, Coppito
  - Research Site, Crema
  - Research Site, Cuneo
  - Research Site, Fano
  - Research Site, Ferrara
  - Research Site, Florence
  - Research Site, Foggia
  - Research Site, Genova
  - Research Site, Iesi
  - Research Site, Latina
  - Research Site, Lecco
  - Research Site, Livorno
  - Research Site, Lugo
  - Research Site, Lungro
  - Research Site, Macerata
  - Research Site, Matera
  - Research Site, Mercatino San Severiono
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Palermo
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Perugia
  - Research Site, Pesaro
  - Research Site, Pescara
  - Research Site, Pietra Ligure
  - Research Site, Pisa
  - Research Site, Pordenone
  - Research Site, Prato
  - Research Site, Reggio Calabria
  - Research Site, Reggio Emilia
  - Research Site, Rocca Priora
  - Research Site, Roma
  - Research Site, Rovigo
  - Research Site, Rozzano
  - Research Site, San Pietro Vernotico
  - Research Site, Sarzana
  - Research Site, Sassari
  - Research Site, Sesto San Giovanni
  - Research Site, Siena
  - Research Site, Syracuse
  - Research Site, Terni
  - Research Site, Torino
  - Research Site, Torrette
  - Research Site, Trapani
  - Research Site, Verona
  - Research Site, Vicenza
  - Research Site, Vimercate
- Netherlands (27):
  - Research Site, 's-Hertogenbosch
  - Research Site, Beek En
  - Research Site, Beerzerveld
  - Research Site, Bennebroek
  - Research Site, Deurne
  - Research Site, Dordrecht
  - Research Site, Echt
  - Research Site, Ermelo
  - Research Site, Fen Haag
  - Research Site, Hoogvliet
  - Research Site, Hoogwoud
  - Research Site, Lieshout
  - Research Site, Losser
  - Research Site, Nijmegen
  - Research Site, Oude Pekela
  - Research Site, Poortvliet
  - Research Site, Rijswijk
  - Research Site, Roelofarends
  - Research Site, Soerendonk
  - Research Site, Spijkenisse
  - Research Site, The Hague
  - Research Site, Voerendaal
  - Research Site, Weerselo
  - Research Site, Wildevank
  - Research Site, Woerden
  - Research Site, Zaandam
  - Research Site, Zutphen
- Norway (12):
  - Research Site, Bergen
  - Research Site, B�verbru
  - Research Site, Elverum
  - Research Site, Fevik
  - Research Site, Fredrikstad
  - Research Site, Larvik
  - Research Site, Løvenstad
  - Research Site, Oslo
  - Research Site, Rådal
  - Research Site, Røa
  - Research Site, Ski
  - Research Site, Ulstet
- Russia (4):
  - Research Site, Kazan’
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Spain (61):
  - Research Site, A Coruña
  - Research Site, Alcalá de Henares
  - Research Site, Alcorcón
  - Research Site, Alicante Orihuela
  - Research Site, Alicante. Elda
  - Research Site, Andújar
  - Research Site, Avilés
  - Research Site, Badajoz
  - Research Site, Bailbao
  - Research Site, Barakaldi/Vizcaya
  - Research Site, Barakaldo Bizkaia
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Cadiz
  - Research Site, Castellon
  - Research Site, Cáceres
  - Research Site, Elche Alicante
  - Research Site, Ferrol
  - Research Site, Fuenlabrada
  - Research Site, Gandia
  - Research Site, Getafe
  - Research Site, Gijón
  - Research Site, Girona
  - Research Site, Granada
  - Research Site, Huelva
  - Research Site, Huercal Overa
  - Research Site, Jaén
  - Research Site, Laredo
  - Research Site, Leganés
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Manacor
  - Research Site, Marbella
  - Research Site, Málaga
  - Research Site, Mérida
  - Research Site, Mostoles Madrid
  - Research Site, Murcia
  - Research Site, Ourense
  - Research Site, Oviedo
  - Research Site, Palencia
  - Research Site, Palma Mallorca
  - Research Site, Pamplona
  - Research Site, Ponferrada
  - Research Site, Pontevedra
  - Research Site, Requena
  - Research Site, Ronda
  - Research Site, Sagunto
  - Research Site, Salamanca
  - Research Site, San Zebastian
  - Research Site, Santa Cruz D E Tenerife
  - Research Site, Santander
  - Research Site, Segovia
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Valladolid
  - Research Site, Viadecans
  - Research Site, Vigo
  - Research Site, Vitoria-Gasteiz
  - Research Site, Vizcaya
  - Research Site, Zaragoza
  - Research Site, Zaroma
- Sweden (29):
  - Research Site, Arvidsjaur
  - Research Site, Åkersberga
  - Research Site, Bromma
  - Research Site, Eskilstuna
  - Research Site, Gävle
  - Research Site, Gothenburg
  - Research Site, Grängesberg
  - Research Site, Hesingborg
  - Research Site, Jarfalla
  - Research Site, Karskrona
  - Research Site, Kil
  - Research Site, Laholm
  - Research Site, Limhamn
  - Research Site, Linköping
  - Research Site, Ludvika
  - Research Site, Luleå
  - Research Site, Malmo
  - Research Site, Nacka
  - Research Site, Örebro
  - Research Site, Piteå
  - Research Site, Stockholm
  - Research Site, Torsås
  - Research Site, Tyreso
  - Research Site, Uppsala
  - Research Site, Vastra Fr�lunda
  - Research Site, Vaxjo
  - Research Site, Vännäs
  - Research Site, Värnamo
  - Research Site, Vinslöv
- United Kingdom (95):
  - Research Site, Airdrie
  - Research Site, Aldershot
  - Research Site, Aylesbury
  - Research Site, Ayrchire
  - Research Site, Barry
  - Research Site, Basildon
  - Research Site, Bath
  - Research Site, Belfast
  - Research Site, Bellshill
  - Research Site, Bexhill-on-Sea
  - Research Site, Blackburn
  - Research Site, Blantyre
  - Research Site, Bolton
  - Research Site, Borehamwood
  - Research Site, Box
  - Research Site, Bracknell
  - Research Site, Bradford-on-Avon
  - Research Site, Burbage
  - Research Site, Bury Saint Edmonds
  - Research Site, Canterbury
  - Research Site, Cardiff
  - Research Site, Chesterfield
  - Research Site, Chippenham
  - Research Site, Coatbridge
  - Research Site, Cookstown
  - Research Site, Corsham
  - Research Site, Coventry
  - Research Site, Crawley
  - Research Site, Crowthorne
  - Research Site, Cumbernauld
  - Research Site, Darlington
  - Research Site, Doncaste
  - Research Site, Dumbarton
  - Research Site, Dumfries
  - Research Site, East Kilbride
  - Research Site, Ecclwsfield
  - Research Site, Ely
  - Research Site, Fowey
  - Research Site, Frome
  - Research Site, Glasgow
  - Research Site, Greenock
  - Research Site, Hamilton
  - Research Site, Headcorn
  - Research Site, High Valleyfield
  - Research Site, Huntington
  - Research Site, Kirkintilloch
  - Research Site, Larne
  - Research Site, Leicester
  - Research Site, Limavady
  - Research Site, Lockerbie
  - Research Site, London
  - Research Site, Maidenhead
  - Research Site, Manhester
  - Research Site, Motherwell
  - Research Site, New Stevenson
  - Research Site, Newcastle
  - Research Site, Newtonstewart
  - Research Site, Newtownabbey
  - Research Site, Northampton
  - Research Site, Norwich
  - Research Site, Nottingham
  - Research Site, Nr Penzance
  - Research Site, Paignton
  - Research Site, Paisley
  - Research Site, Penzance
  - Research Site, Peterborough
  - Research Site, Plymouth
  - Research Site, Port Glasgow
  - Research Site, Praze-on-Beeble
  - Research Site, Reading
  - Research Site, Redditch
  - Research Site, Renfrew
  - Research Site, Saltash
  - Research Site, Sandy
  - Research Site, Sheffield
  - Research Site, Shepshed
  - Research Site, Slough
  - Research Site, Spalding
  - Research Site, Spennymoor
  - Research Site, Strathaven
  - Research Site, Strathblane
  - Research Site, Sunbury-on-Thames
  - Research Site, Swindon
  - Research Site, Thornhill
  - Research Site, Thornton Heath
  - Research Site, Tichfield
  - Research Site, Torpoint
  - Research Site, Trowbridge
  - Research Site, Walsall
  - Research Site, Welingborough
  - Research Site, Wells-next-the-Sea
  - Research Site, Weston-super-Mare
  - Research Site, Whitstable
  - Research Site, Wishaw
  - Research Site, Yaxley

REFERENCES:
- [Derived] Aubier M, Haughney J, Selroos O, van Schayck OC, Ekstrom T, Ostinelli J, Buhl R. Is the patient's baseline inhaled steroid dose a factor for choosing the budesonide/formoterol maintenance and reliever therapy regimen? Ther Adv Respir Dis. 2011 Oct;5(5):289-98. doi: 10.1177/1753465811407236. Epub 2011 May 17. PMID 21586508
- [Derived] Haughney J, Aubier M, Jorgensen L, Ostinelli J, Selroos O, van Schayck CP, Buhl R. Comparing asthma treatment in elderly versus younger patients. Respir Med. 2011 Jun;105(6):838-45. doi: 10.1016/j.rmed.2011.02.011. Epub 2011 Mar 23. PMID 21435854
- [Derived] Aubier M, Buhl R, Ekstrom T, Ostinelli J, van Schayck CP, Selroos O, Haughney J. Comparison of two twice-daily doses of budesonide/formoterol maintenance and reliever therapy. Eur Respir J. 2010 Sep;36(3):524-30. doi: 10.1183/09031936.00022010. Epub 2010 Jul 1. PMID 20595145

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 6-month, randomised, open label, parallel-group, active controlled, multinational study, in participants with uncontrolled/partly controlled asthma, who were symptomatic despite daily use of inhaled glucocorticosteroid (IGCS) with or without Long-Acting β2 agonist (LABA).
Groups:
- Symbicort® SMART®) 1*2: 1 inhalation of Symbicort 160µg/4.5µg twice daily plus as-needed.
- Symbicort® SMART®) 2*2: 2 inhalations of Symbicort 160µg/4.5µg twice daily plus as-needed.
Period: Overall Study
Arm/Group | Symbicort® SMART®) 1*2 | Symbicort® SMART®) 2*2
Started | 4008 (4203 participants randomised. Out of these, 195 had no efficacy data after randomisation.) | 4045 (4221 participants randomised. Out of these, 176 had no efficacy data after randomisation.)
Completed | 3699 | 3705
Not Completed | 309 | 340
Not completed — Adverse Event | 70 | 93
Not completed — Withdrawal by Subject | 81 | 79
Not completed — Lost to Follow-up | 46 | 55
Not completed — Incorrect Enrolment | 64 | 66
Not completed — Severe Non-Compliance to Protocol | 25 | 21
Not completed — Safety Reason | 1 | 3
Not completed — Mis-Randomization of subject | 0 | 1
Not completed — Other | 22 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort® SMART®) 1*2 | Symbicort® SMART®) 2*2 | Total
Number analyzed (Participants) | 4008 | 4045 | 8053
Age Continuous [Mean (Full Range); unit: Years] | 47.8 [18 to 96] | 47.9 [18 to 90] | 47.8 [18 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2483 | 2512 | 4995
  Male | 1525 | 1533 | 3058
Treatment with Long-Acting β2 agonist (LABA) at baseline. [Number; unit: Participants]
  Number of participants using LABA at baseline. | 3108 | 3118 | 6226
  Number of participants without LABA at baseline. | 900 | 927 | 1827
Asthma control questionnaire (ACQ5) score at study entry [Mean (Standard Deviation); unit: Units on a scale] — ACQ5 was used. The lower value the better with a full range from 0=no impairment, 6= maximum impairment. Awakenings, morning symptoms, limitations, shortness of breath and wheeze.
  Units on a scale
    ACQ5 score at study entry | 1.85 (0.98) | 1.86 (1.01) | 1.85 (0.99)
Exacerbations past 12 months before study start. [Mean (Standard Deviation); unit: Number of exacerbations per participant] | 1.47 (2.42) | 1.42 (2.42) | 1.45 (2.42)
Inhaled glucocorticosteroids (IGCS) dose at study entry. [Mean (Standard Deviation); unit: μg/day]
  IGCS dose at study entry | 1046 (595) | 1037 (575) | 1042 (585)
Participants with a well controlled asthma week at study entry. [Mean (Full Range); unit: Percentage of participants] | 11.97 [0 to 100] | 11.77 [0 to 100] | 11.87 [0 to 100]
Pulmonary function test at baseline. [Mean (Full Range); unit: Percent of predicted normal value of PEF] — Peak Expiratory Flow (PEF) was recorded at baseline, the assessment was performed at least 15 minutes after 2 inhalations of Symbicort 160/4.5µg. pn=predicted normal. Symbicort SMART 1*2 arm: n=4001 and Symbicort SMART 2*2 arm: n=4003.
  Percent of predicted normal value of PEF
    Percent Included | 90.8 [0 to 100] | 90.1 [0 to 100] | 90.4 [0 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Number of Severe Asthma Exacerbations Per Participant.
Description: Time to first severe asthma exacerbation, translated to mean number of severe asthma exacerbations per participant. A severe asthma exacerbation is defined as deterioration in asthma requiring oral/systemic glucocorticosteroids for at least 3 days and/or hospitalisation/emergency room visit with oral/systemic glucocorticosteroid treatment.
Time Frame: 6 months
Measure: Mean (Full Range); unit: Severe exacerbations per participant
Arm/Group | Symbicort® SMART®) 1*2 | Symbicort® SMART®) 2*2
Number analyzed (Participants) | 4008 | 4045
Severe exacerbations per participant | 0.097 (0) [0 to 4] | 0.080 (0) [0 to 5]

2. Secondary Outcome: Fraction of Participants With Severe Asthma Exacerbation
Description: The total number of severe asthma exacerbations was calculated for each participant. A severe asthma exacerbation is defined as deterioration in asthma requiring oral/systemic glucocorticosteroids for at least 3 days and/or hospitalisation/emergency room visit with oral/systemic glucocorticosteroid treatment.
Time Frame: 6 months.
Measure: Mean (95% Confidence Interval); unit: Fraction of participants with event
Arm/Group | Symbicort® SMART®) 1*2 | Symbicort® SMART®) 2*2
Number analyzed (Participants) | 4008 | 4045
Fraction of participants with event | 0.09686 (0.08528) [0.08528 to 0.11] | 0.07955 (0.06927) [0.06927 to 0.09135]

3. Secondary Outcome: Total Number of Severe Asthma Exacerbations That Led to Hospitalisation and/or Emergency Room Treatment.
Description: A severe asthma exacerbation is defined as deterioration in asthma requiring oral/systemic glucocorticosteroids for at least 3 days and/or hospitalisation/emergency room visit with oral/systemic glucocorticosteroid treatment. Number of events per participant
Time Frame: 6 months.
Measure: Mean (Full Range); unit: Number of events per participant
Arm/Group | Symbicort® SMART®) 1*2 | Symbicort® SMART®) 2*2
Number analyzed (Participants) | 4008 | 4045
Number of events per participant | 0.0120 (0) [0 to 3] | 0.0091 (0) [0 to 2]

4. Secondary Outcome: Total Number of Days Per Participant With Oral/Systemic Glucocorticosteroids During Severe Asthma Exacerbation
Description: Total number of days with oral/systemic glucocorticosteroids during severe exacerbation calculated for each participant. A severe asthma exacerbation is defined as deterioration in asthma requiring oral/systemic glucocorticosteroids for at least 3 days and/or hospitalisation/emergency room visit with oral/systemic glucocorticosteroid treatment.
Time Frame: 6 months.
Measure: Mean (Standard Deviation); unit: Days per participant
Arm/Group | Symbicort® SMART®) 1*2 | Symbicort® SMART®) 2*2
Number analyzed (Participants) | 4008 | 4045
Days per participant | 9.6 (8.1) | 9.1 (5.5)

5. Secondary Outcome: Mean Daily Number of Inhalations of As-needed Medication.
Description: The number of as-needed inhalations was measured 2 times during 2 weeks before 13 weeks and 26 weeks of treatment.
Time Frame: 4 weeks
Population: Inhalations of as-needed medication recorded by 3880 participants in the Symbicort SMART 1*2 Reporting Group and recorded by 3881 participants in the Symbicort SMART 2*2 Reporting Group
Measure: Mean (Full Range); unit: Inhalations per day per participant
Arm/Group | Symbicort® SMART®) 1*2 | Symbicort® SMART®) 2*2
Number analyzed (Participants) | 3880 | 3881
Inhalations per day per participant | 0.897 (0) [0 to 9.14] | 0.625 (0) [0 to 9.07]

6. Secondary Outcome: Percent of Participants With a Well Controlled Asthma Week.
Description: The mean percent of participants fulfilling the criteria for a well controlled asthma week in each treatment. A well controlled asthma week is defined as a week with no exacerbations and no night-time awakenings due to asthma and a maximum of 2 days with symptoms and as-needed inhalation use.
Time Frame: 6 months.
Population: Data for this measure recorded by 3714 participants in the Symbicort SMART 1*2 Reporting Group and recorded by 3718 participants in the Symbicort SMART 2*2 Reporting Group.
Measure: Mean (Full Range); unit: Percentage of participants
Arm/Group | Symbicort® SMART®) 1*2 | Symbicort® SMART®) 2*2
Number analyzed (Participants) | 3714 | 3718
Percentage of participants | 43.69 (0) [0 to 100] | 54.26 (0) [0 to 100]

7. Secondary Outcome: Mean Overall Asthma Control Questionnaire (ACQ) Score
Description: The ACQ5 was used. The lower value the better with a full range from 0=no impairment, 6= maximum impairment. Awakenings, morning symptoms, limitations, shortness of breath and wheeze.
Time Frame: 6 months.
Population: Data for this measure recorded by 3709 participants in the Symbicort SMART 1*2 Reporting Group and recorded by 3735 participants in the Symbicort SMART 2*2 Reporting Group.
Measure: Mean (Full Range); unit: Scores in a scale
Arm/Group | Symbicort® SMART®) 1*2 | Symbicort® SMART®) 2*2
Number analyzed (Participants) | 3709 | 3735
Scores in a scale | 1.18 (0) [0 to 5.7] | 1.089 (0) [0 to 5.0]

8. Secondary Outcome: The Mean Total Daily Dose of Steroids From Symbicort.
Description: The mean total daily dose of steroids from Symbicort was calculated as the sum of the maintenance dose and the as-needed dose.
Time Frame: 4 weeks
Population: : Data for this measure recorded by 3874 participants in the Symbicort SMART 1*2 Reporting Group and recorded by 3873 participants in the Symbicort SMART 2*2 Reporting Group.
Measure: Mean (Standard Deviation); unit: μg budesonide per day
Arm/Group | Symbicort® SMART®) 1*2 | Symbicort® SMART®) 2*2
Number analyzed (Participants) | 3874 | 3873
μg budesonide per day | 462.96 (179.10) | 736.58 (152.70)

9. Secondary Outcome: Mean Cost Per Participant Per Country
Description: Mean cost is calculated for each country using participants from the whole study and country specific costs. Mean value for the whole study can not be calculated.
Time Frame: 6 months
Reporting Status: Not Posted
Measure: Mean (Full Range); unit: Euro

ADVERSE EVENTS:
Arm/Group | Symbicort® SMART®) 1*2 | Symbicort® SMART®) 2*2
Serious Adverse Events (participants affected / at risk) | 77/4008 | 88/4045
Other Adverse Events (participants affected / at risk) | 0/4008 | 0/4045
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort® SMART®) 1*2 (N=4008) | Symbicort® SMART®) 2*2 (N=4045)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Angina Pectoris (Cardiac disorders) | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 1
Atrioventricular Block (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Exomphalos (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Crohn's Disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Diverticulum Intestinal (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Reflux Oesophagitis (Gastrointestinal disorders) | 1 | 0
Salivary Gland Enlargement (Gastrointestinal disorders) | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 2 | 1
Cyst (General disorders) | 0 | 1
Death (General disorders) | 1 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 4
Food Allergy (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
Bronchiectasis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2
Campylobacter Gastroenteritis (Infections and infestations) | 1 | 0
Chronic Sinusitis (Infections and infestations) | 0 | 1
Epstein-Barr Virus Infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 1
Lung Infection (Infections and infestations) | 0 | 1
Meningitis Viral (Infections and infestations) | 0 | 1
Pilonidal Cyst (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 3
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Animal Bite (Injury, poisoning and procedural complications) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 2
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 | 0
Multiple Drug Overdose (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle Mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 3
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Vocal Cord Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid Sinus Syndrome (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 2
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic Stroke (Nervous system disorders) | 1 | 0
Ischaemic Cerebral Infarction (Nervous system disorders) | 1 | 0
Loss Of Consciousness (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other